CLINICAL TRIAL: NCT06092112
Title: A Clinical Trial for the Safety and Efficacy of CD-801 in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital,, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-HCC-2023-IIT-EX
Record Dates: First submitted 2023-10-07; First posted 2023-10-23 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; HNF4α
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The subjects with advanced HCC will be treated by CD-801 through the hepatic artery injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-801 treatment (Experimental): The subjects with advanced HCC will be treated by CD-801 through the hepatic artery injection.
  Interventions: Drug: CD-801

INTERVENTIONS:
Drug: CD-801 — The subjects with advanced HCC will be treated by 100 μg CD-801 through the hepatic artery injection at two-week intervals. The dosing interval will be adjusted based on subject tolerability, safety, and efficacy. For example, it may be adjusted to administer the medication once every three weeks or four weeks.

SUMMARY:
The goal of this investigator-initiated, a single-arm, open-label, pilot study is to investigate the safety, tolerability, and efficacy of CD-801 treatment in subjects with advanced hepatocellular carcinoma.

Condition of disease: advanced hepatocellular carcinoma .

Intervention：treatment with 100μg CD-801 through the hepatic artery at two-week intervals. The dosing interval will be adjusted based on subject tolerability, safety, and efficacy. For example, it may be adjusted to administer the medication once every three weeks or four weeks.

Drug: CD-801, a drug designed specifically to enhance the expression of HNF4α and selectively target liver cancer cells.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common form of liver cancer. Recent advancements in understanding tumor biology and the tumor microenvironment have dramatically transformed the treatment landscape for advanced stage HCC. However, the survival for advanced HCC patients still remains unsatisfactory.

Differentiation therapy in oncology is defined as a therapeutic strategy that reactivates endogenous differentiation programs and reverts malignant phenotypes. Its hallmark success is the treatment of acute promyelocytic leukemia (APL) by the combination of all-trans retinoic acid (ATRA) and arsenic. Unfortunately, this approach has achieved limited success in solid tumors.

Hepatocyte nuclear factor 4α (HNF4α) is a transcription factor (TF) belonging to the nuclear receptor family. HNF4α is highly enriched in mature hepatocytes and serves as a master regulator of hepatocyte differentiation and hepatic metabolism. Previous studies, including the investigators' and others, have demonstrated that the reduced expression of HNF4α plays a critical role in hepatocarcinogenesis. Restoring HNF4α expression induces the differentiation of HCC cells into mature hepatocytes and has shown significant therapeutic effects in various animal models of HCC.

In this study, the investigators developed CD-801, a drug designed specifically to enhance the expression of HNF4α and selectively target liver cancer cells, for the treatment of HCC patients. Preclinical studies have shown that CD-801 effectively inhibits the growth of subcutaneous and orthotopic liver tumors in mice. Acute toxicity tests in SD rats have demonstrated that a single intravenous injection of CD-801 injection at a dose of 150 μg/animal is well-tolerated, with no significant toxicity, indicating good safety profiles. Furthermore, in the dose escalation phase of the clinical trial which the investigators have completed, CD-801(25, 50 and 100 μg) was found to be well-tolerated. None of the patients experienced dose-limiting toxicities (DLTs) during the DLT phase.

This trial is a single-arm, open-label, exploratory clinical study aimed at further evaluating the efficacy, safety, and tolerability of 100 μg CD-801 administered through the hepatic artery in the treatment of advanced-stage HCC at two-week intervals (The dosing interval will be adjusted based on subject tolerability, safety, and efficacy. For example, it may be adjusted to administer the medication once every three weeks or four weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older.
2. Subjects must have confirmed diagnosis of HCC according to the American Association for the Study of Liver Diseases criteria.
3. Unresectable HCC.
4. Subjects are unsuitable for local or systemic anti-tumor therapy or had tumor progression after receiving at least one kind of conventional treatment.
5. According to mRECIST, subjects should be with at least 1 measurable target lesion.
6. Life expectancy of 12 weeks or more.
7. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
8. Male with fertility and females of childbearing potential are willing to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation. Females of childbearing age, including premenopausal females and within 2 years after menopause, must have a negative serum pregnancy test result within 7 days prior to the first dose of study treatment.
9. Subjects who have voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. ALB < 28 g/L, or Bilirubin >5.0 mg/dL, or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) >5×ULN.
2. Inadequate renal function defined as creatinine >1.5 times the upper limit of normal (ULN) or calculated creatinine clearance < 40 mL/min.
3. Absolute neutrophil count (ANC) < 1.0×109/L, or Platelets < 30×109/L, or Hemoglobin < 8.5 g/dL.
4. International Normalized Ratio (INR) > 2.3.
5. Subjects with a history of liver transplantation.
6. Subjects with poorly controlled hypertension, diabetes or other serious heart or lung diseases, or with serious dysfunction.
7. Subjects with extrahepatic metastasis who had potential benefit from first-line systemic therapies.
8. Subjects who had prior anticancer treatment with any locoregional therapies, antiangiogenic targeted therapies, immune checkpoint inhibitors or chemotherapy within 4 weeks (within 2 weeks in case of sorafenib), radiotherapy within 3 weeks, or active traditional Chinese medicine within 2 weeks before the first dose of study treatment, except for the treatments after which the disease still progressed according to mRECIST.
9. All toxicities related to prior locoregional or systemic anti-tumor treatments are still grade 2 or more (except for hair loss and other events that have been judged tolerable by researchers).
10. Subjects with complication histories of liver cirrhosis or HCC such as gastrointestinal hemorrhage, overt hepatic encephalopathy, or uncontrollable ascites within 2 weeks prior to the first dose of study treatment.
11. Uncontrolled active infection (eg, lung infections, or abdominal infections).
12. Subjects with moderate to severe hepatic artery- portal vein fistula or hepatic artery - vein fistula which could not be avoided even through the artery super selection by DSA.
13. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated early gastric carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or localized prostate cancer.
14. HBV DNA greater than 500 copies/mL, or HCV RNA greater than 15 U/mL.
15. Subject is positive for Human Immunodeficiency Virus (HIV).
16. Any subject who is allergic to MRI contrast agents.
17. Pregnant/lactating women, or women who have the possibility of pregnancy.
18. Participation in other investigational drug trials within 4 weeks prior to initiation of this study treatment.
19. Any medical or other condition which, in the opinion of the investigator, would preclude participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
The objective response rate based on mRECIST | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on mRECIST

SECONDARY OUTCOMES:
Adverse events as assessed by CTCAE v5.0 | Through study completion, an average of 2 years
  To assess the incidence and severity of AE after CD-801 treatment in subjects with advanced hepatocellular carcinoma by CTCAE v5.0
The objective response rate based on RECIST v1.1 | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on RECIST v1.1
Duration of response based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first documentation of complete response or partial response to the date of first documentation of disease progression or death (whichever occurs first) based on mRECIST and RECIST v1.1
Progression-free survival based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurs first) based on mRECIST and RECIST v1.1
Time to progression based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression based on mRECIST and RECIST v1.1
Time to response based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the date of first study dose to the date of first documentation of complete response or partial response based on mRECIST and RECIST v1.1
Disease control rate based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or stable disease (minimum duration from C1D1 to stable disease ≥5 weeks) based on mRECIST and RECIST v1.1
Clinical benefit rate based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or durable stable disease (duration of stable disease ≥ 23 weeks) based on mRECIST and RECIST v1.1
Overall Survival | Throughout the entire course of treatment until the end of the follow-up period, an average of 2 years
  To assess the time from the first study dose date until date of death from any cause . Subjects who are lost to follow-up and the subjects who are alive at the date of data cutoff will be censored at the date the subject was last known alive or the cut-off date, whichever comes earlier.

OTHER OUTCOMES:
Health Related Quality of Life based on the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30. | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30.
Health Related Quality of Life based on HCC-specific EORTC QLQ-HCC18 questionnaire. | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using HCC-specific EORTC QLQ-HCC18 questionnaire.
Health Related Quality of Life based on European Quality of Life questionnaire. | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using European Quality of Life questionnaire.
The impact of CD-801 treatment on cytokine in serum after treatment. | Through study completion, an average of 2 years
  To investigate the changes of cytokine in serum in subjects with advanced hepatocellular carcinoma after CD-801 treatment
The impact of CD-801 treatment on immune cell profiling in serum after treatment. | Through study completion, an average of 2 years
  To investigate the changes of immune cell profiling in serum in subjects with advanced hepatocellular carcinoma after CD-801 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, M.D., Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Changzheng Hospital，Naval Medical University, Shanghai, Shanghai Municipality, China